CLINICAL TRIAL: NCT06926907
Title: Development and Evaluation of the T.E.A.C.H. Study: A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Principal Investigator, Catherine Coccia, PhD, RD, Associate Professor, Florida International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-22-0373
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Child Obesity
Keywords: Teacher intervention; Montessori schools; Obesity Prevention; Nutrition education; Randomized control trial
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: This study employed a cluster randomized waitlist control design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants in this arm received the 6-week online T.E.A.C.H. program.
  Interventions: Behavioral: The Teacher Education and Classroom Habits (T.E.A.C.H.) Program
- Control (No Intervention)

INTERVENTIONS:
Behavioral: The Teacher Education and Classroom Habits (T.E.A.C.H.) Program — The T.E.A.C.H. Program utilized essential constructs of the Social Cognitive Theory to deliver virtual nutrition education to Montessori teachers over a 6-week period. The intervention consisted of four program components: 1. An interactive online nutrition education platform with 6 modules was developed using a WordPress website. Each module contained 5 topics including adult nutrition, child nutrition, classroom food practices, cultural practices, and teacher-parent communication. Teachers were provided login information via email containing a unique identifier to be used as their username and were prompted to complete one module per week for 6 weeks; 2. Live weekly virtual education sessions were held via Zoom to supplement and reinforce the online learning experience; 3. A Montessori-based nutrition curriculum with 6 weekly lessons to utilize in the classroom was provided to each participant; 4. Educational handouts to be disseminated to parents.
  Arms: Intervention

SUMMARY:
Using a randomized control design, this study seeks to develop and evaluate a nutrition intervention to increase Montessori teachers' nutrition knowledge, nutrition self-efficacy, nutrition teaching self-efficacy and cultural food competence to improve teachers' eating behaviors, nutrition teaching practices, classroom food practices, and teacher-parent communication. This study will examine the feasibility and efficacy of a nutrition intervention for teachers which will include a nutrition education program via an online platform and hands-on Montessori-based curriculum to teach nutrition in the classroom. Teachers from multiple schools will be recruited using the public national Montessori listserv. This study will enhance teachers' nutrition knowledge which may increase their nutrition teaching practices and improve their personal nutrition habits. Improving teachers' personal and classroom nutrition practices may improve teachers' personal health outcomes and may positively impact their students through modeling of healthy behaviors and improving the classroom food environment.

ELIGIBILITY:
Inclusion Criteria:

Teachers were considered eligible to participate in the study if they taught in early childhood classrooms (students 3 to 6 years old), were ≥ 18 years old, and had access to an electronic device with internet connection and audiovisual capabilities.

Exclusion Criteria:

Teachers were deemed ineligible to participate if they were not fluent in English (written & verbal) or had plans to leave their place of employment during the study timeframe

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the mean Nutrition Knowledge at 12 week follow-up | From enrollment to the end of the 12 week follow-up.
  Teachers' nutrition knowledge was measured using subscales 1 and 2 from the revised General Nutrition Knowledge Questionnaire (GNKQ-R).
Change from Baseline in the mean Nutrition Self-efficacy at 12 week follow-up | From enrollment to the end of the 12 week follow-up.
  Nutrition self-efficacy was determined using the Dewar's Nutrition Self-Efficacy Scale.
Change from Baseline in the mean Nutrition teaching self-efficacy at 12 week follow-up | From enrollment to the end of the 12 week follow-up.
  Nutrition teaching self-efficacy was determined using the Nutrition Teaching Self-Efficacy Scale.
Change from Baseline in the mean cultural competence at 12 week follow-up | From enrollment to the end of the 12 week follow-up.
  The Multicultural Teaching Competency Scale Teachers' was utilized to measure teachers' cultural competence.

SECONDARY OUTCOMES:
Change from Baseline in the mean classroom eating behaviors at 12 week follow-up | From enrollment to the end of the 12 week follow-up.
  Teachers' eating behaviors were measured using the Teacher's Classroom Eating Behaviors tool
Change from Baseline in the mean classroom food practices at 12 week follow-up | From enrollment to the end of the 12 week follow-up.
  Classroom food practices were determined using Classroom Food-Related Practices-to-Limit Scale.
Change from Baseline in the mean nutrition teaching practices at 12 week follow-up | From enrollment to the end of the 12 week follow-up.
  Subscale 2 of the Nutrition Education Practices (NEP) Survey for Teachers and Foodservice Directors was utilized to measure nutrition teaching practices.
Change from Baseline in the mean teacher-parent nutrition communication at 12 week follow-up | From enrollment to the end of the 12 week follow-up.
  Teachers' communication with parents was measured using subscale 2 of the Teacher-Parent Contact Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No